CLINICAL TRIAL: NCT06354543
Title: Safety and Clinical Performance Assessment of Bone Cements and Cement Restrictor Used in Arthroplasty - A Post-market Clinical Follow-up
Brief Title: Arthroplasty Cements Outcomes - A Post-market Follow-up
Status: Recruiting | Type: Observational
Sponsor: Teknimed (Industry)
Responsible Party: Sponsor
Other Study IDs: CA01-TK-ARTHRO
Record Dates: First submitted 2024-03-22; First posted 2024-04-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Arthroplasty
Keywords: cement; prosthesis; arthroplasty; knee; hip; shoulder; joint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (21):
- CEMFIX1 Knee primary surgery: Patients included for primary knee surgery with CEMFIX 1
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX1 Knee revision surgery: Patients included for revision knee surgery with CEMFIX 1
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX1 Hip primary surgery: Patients included for primary hip surgery with CEMFIX 1
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX1 Hip revision surgery: Patients included for revision hip surgery with CEMFIX 1
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX1 Shoulder primary surgery: Patients included for primary shoulder surgery with CEMFIX 1
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX1 Shoulder revision surgery: Patients included for revision shoulder surgery with CEMFIX 1
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX3 Hip primary surgery: Patients included for primary hip surgery with CEMFIX 3
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX3 Hip revision surgery: Patients included for revision hip surgery with CEMFIX 3
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX3 Shoulder primary surgery: Patients included for primary shoulder surgery with CEMFIX 3
  Interventions: Device: Cemented joint arthroplasty
- CEMFIX3 Shoulder revision surgery: Patients included for revision shoulder surgery with CEMFIX 3
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX1 Knee primary surgery: Patients included for primary knee surgery with GENTAFIX 1
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX1 Knee revision surgery: Patients included for revision knee surgery with GENTAFIX 1
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX1 Hip primary surgery: Patients included for primary hip surgery with GENTAFIX 1
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX1 Shoulder primary surgery: Patients included for primary shoulder surgery with GENTAFIX 1
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX3MV Hip primary surgery: Patients included for primary hip surgery with GENTAFIX 3MV
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX3MV Hip revision surgery: Patients included for revision hip surgery with GENTAFIX 3MV
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX3MV Knee revision surgery: Patients included for revision knee surgery with GENTAFIX 3MV
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX3 Knee revision surgery: Patients included for revision knee surgery with GENTAFIX 3
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX3 Hip primary surgery: Patients included for primary hip surgery with GENTAFIX 3
  Interventions: Device: Cemented joint arthroplasty
- GENTAFIX3 Hip revision surgery: Patients included for revision hip surgery with GENTAFIX 3
  Interventions: Device: Cemented joint arthroplasty
- CEMSTOP Hip surgery: Patients included for hip surgery with CEMSTOP
  Interventions: Device: Cemented joint arthroplasty

INTERVENTIONS:
Device: Cemented joint arthroplasty — Joint replacement with cemented prosthetic components

SUMMARY:
A Post-Market Clinical Follow-Up (PMCF) Study to collect clinical data on safety and performance of all Teknimed Arthroplasty range of products: CEMFIX® and GENTAFIX® bone cements families and CEMSTOP® cement restrictor, and all their private labels.

Teknimed bone cements and cement restrictor are legacy products, some marketed for more than 20 years. Their performance and safety have already been demonstrated by Post-Market Surveillance and previous clinical studies. The current Post-Market Clinical Follow-Up study aims to confirm these claims by collecting data in a "real-life" setting.

The study is a retrospective and prospective global, single arm, non-controlled, multicentric, ambispective observational study. Patients will be followed as per local standard medical care of the site.

DETAILED DESCRIPTION:
It is admitted that:

* Joint replacement is a commonly performed major surgical procedure that has considerable success in alleviating pain and disability;
* These procedures may be done with the help of a bone cement (PMMA) to fix the prosthesis to the bone (cemented fixation);
* Most common reasons for primary joint replacement are osteoarthritis, osteonecrosis and trauma;
* Most common reasons for revision of joint replacement are dislocation, infection, fracture and prothesis loosening;
* Quality of bone cement have a large influence on long-term implant stability.

TEKNIMED has developed several bone cements and a cement restrictor currently used in arthroplasty procedures.

With the increasing use of these procedures, there is a need of real-life long-term safety and efficacy data on the bone cements.

This retro- and prospective study is performed to assess the safety and performance of TEKNIMED arthroplasty products in their current clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Be willing to sign an informed consent approved by Institutional Review Board (IRB) or European Commission (EC) (when applicable) or not oppose to the use of their clinical data in the study
* For prospective inclusion: be considered for an arthroplasty procedure with one of the TEKNIMED orthopaedic cement and/or cement restrictor comprised in this study (primary or revision surgery).
* For retrospective inclusion: have undergone a primary or revision arthroplasty procedure with a TEKNIMED orthopaedic cement and/or cement restrictor between the 1st January 2016 and the date of the site initiation visit (SIV).
* Be informed of the study and not being opposed to the use of their clinical data in the study or be willing to sign an informed consent during the first follow-up visit following the site initiation (where applicable).

Exclusion Criteria:

* Patient under trusteeship or guardianship,
* Women who are pregnant
* Patient unable to follow the protocol
* Patient whose vital prognosis is unfavorable (according to investigator's opinion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for whom a cemented arthroplasty surgery is indicated
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 15 years (until the lifetime of the device)
  Prosthesis survival defined as time from implantation to revision surgery due to a cement defect.
Superficial and/or deep postoperative infection rate. | 15 years (until the lifetime of the device)
  In the case of cements with gentamicin, superficial and/or deep postoperative infection rate.

SECONDARY OUTCOMES:
Pain Level | 5 years
  Pain evaluated by Visual Analogue Scale (VAS): on a scale of 0 to 10, with 0 being no pain and 10 being the most severe pain at the Baseline and at the Follow-up visits
Patients' satisfaction | 5 years
  Patient satisfaction assessed using a 3-question patient satisfaction questionnaire (Yes/No/Without opinion) at the Follow-up visits
Restoration of function | 5 years
  Evaluation of mobility by functional scores: "Constant Score" for the shoulder (scale of 100 points, 100 points is the best mobility) at the baseline and at the Follow-up visits
Evaluation of function and radiological outcomes | 5 years
  "SEDEL Score" at the Follow-up visits ( A: no pejorative functional and radiographic signs / B: patients with stable clinical result but demonstrating progressively evolving radiographic alterations / C: patients with deteriorating functional score but lack of any radiographic explanation / D: patients with bad clinical score associated with progressive radiographic deterioration)
Complications rate | 5 years
  Evaluation of complications will be assessed on radiological images: cement leakage, implant migration, radiolucent lines, osteolytic zone at the Follow-up visits
Antalgic consumption | 5 years
  Antalgic consumption and the drug type at the Baseline and at the Follow-up visits
Restoration of function | 5 years
  Evaluation of mobility by functional scores: "Postel Merle d'Aubigne score" (PMA) for the hip (scale of 18 points, 18 points is the best functional score) at the Baseline and at the Follow-up visits
Restoration of function | 5 years
  Evaluation of mobility by functional scores: "Tegner Lysholm Knee Score" for the knee (scale of 100 points, 100 points is the best functional score) at the Baseline and at the Follow-up visits
Adverse events | 15 years (until the lifetime of the device)
  All adverse events (such as prosthesis loosening rate, dislocation, deep infection …) occured during surgery and through study completion

CONTACTS AND LOCATIONS:
Locations (10):
- France (8):
  - CH de Brive, Brive-la-Gaillarde, Aquitaine
  - Clinique du Vivarais, Aubenas, Auvergne-Rhône-Alpes
  - Clinique du Val d'Ouest, Écully, Auvergne-Rhône-Alpes
  - Cabinet de consultation, Évreux, Eure
  - Clinique du Dr Henri Guillard, Coutances, Normandy
  - Clinique de l'Atlantique, Puilboreau, Nouvelle-Aquitaine
  - MIROUSE, Boujan-sur-Libron, Occitanie
  - Hôpital Européen Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
- Italy (2):
  - Instituto Ortopedico Rizzoli, Bologna, Emilia-Romagna
  - Ospedale Santissima Annunziata, Cento, Emilia-Romagna

IPD SHARING:
Plan to Share IPD: No